CLINICAL TRIAL: NCT01100580
Title: The Links Between Water and Salt Intake, Body Weight, Hypertension and Kidney Stones: a Difficult Puzzle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Parma (Other)
Responsible Party: Prof. Loris Borghi, University of Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORST-1028
Record Dates: First submitted 2010-03-29; First posted 2010-04-09 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Urinary Stones; Hypertension; Overweight; Obesity
Keywords: Low-salt diet; calciuria; blood pressure; nephrolithiasis; hypertension; BMI; urinary stone risk factors
MeSH Terms: conditions — Urinary Calculi; Hypertension; Overweight; Obesity; Nephrolithiasis | interventions — Diet, Sodium-Restricted; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- water therapy (Active Comparator): The term "water therapy" refers to an abundant intake of water with a low mineral and low sodium content (at least 2 litres in winter and 3 in summer).
  Interventions: Dietary Supplement: water therapy
- low salt diet + water therapy (Experimental): low salt diet refers to a salt intake of 4 g/day
  Interventions: Dietary Supplement: low salt diet

INTERVENTIONS:
Dietary Supplement: low salt diet — Daily salt intake less than 4 g/day
  Arms: low salt diet + water therapy
Dietary Supplement: water therapy — abundant intake of water with a low mineral and low sodium content (at least 2 litres in winter and 3 in summer).
  Arms: water therapy

SUMMARY:
Nephrolithiasis is a disease that strikes roughly 10% of the Italian population and its incidence in industrialized countries is on the increase. The most common form of the disease (80%) is Idiopathic Calcium Nephrolithiasis (ICN) with calcium-oxalate (CaOx) and/or calcium-phosphate (CaP) stones. The etiopathogenesis involves both genetic and acquired factors, the interplay of which leads to urinary biochemical anomalies at the root of stone formation. The elements and urinary compounds involved are known as "urinary stone risk factors". The risk factors for CaOx stones consist of low urine volume, hypercalciuria, hyperoxaluria, hyperuricosuria, hypocitraturia and hypomagnesuria. In the case of CaP stones, the hyperphosphaturia and pH parameters are of particular importance; a pH>7 promotes the formation of stones prevalently composed of phosphates, while a pH of between 6 and 7, associated with a volume <1l/day, can raise CaP supersaturation to a dangerously high level and lead to the formation of mixed CaOx and CaP stones. For uric acid stones, the elements involved are hyperuricosuria and pH<5.5. In general, the most prevalent alteration in ICN is hypercalciuria (50%). Hypertension and obesity are also social diseases with important epidemiological similarities to nephrolithiasis. These affinities have led to the search for a common pathogenic moment. As far as hypertension is concerned, various studies have demonstrated high calciuria in hypertensives with a linear relationship between 24-h calciuria and arterial blood pressure. The incidence of stone disease is greater in hypertensives than in normotensives and, by the same token, the incidence of hypertension is greater in stone formers than in non stone formers, but it is not clear whether nephrolithiasis is a risk factor for hypertension or vice versa. Moreover, a linear relationship exists between calciuria and natriuria, where the calcium is the dependent variable, with a much steeper slope of the straight line in stone formers and hypertensives compared to controls. It has, in fact, been demonstrated that to reduce calcium, it is more efficacious to reduce sodium intake as opposed to calcium intake. Finally, BMI and body weight are independently associated with an increase in stone risk even though, due to a number of bias (limited weight categories, low number of obese persons in the study populations, no control group, no recording of food intake) the studies published failed to be conclusive. In the final analysis, stone disease, arterial hypertension and excess weight/obesity prove to be closely interconnected and it is possible to intervene with targeted diets aimed at reducing the risk of illness and death from these diseases. Among such dietary approaches, the reduction of sodium chloride in food, increased hydration and an increased intake of foods with an alkaline potential seem to play an important role.

For many years now, the investigators research unit has been involved in projects, partially financed by the Italian Ministry of University and Research (MIUR), geared towards studying the effects induced by dietary changes in patients with calcium stone disease. The aim of the present project is to analyse in depth the relationship between stone disease, hypertension, body weight and water and salt intake both in the general population of the area of Parma (where historically and by gastronomic tradition, the usual diet tends to have a high salt content) and in a selected population of stone formers and hypertensives not under treatment. A representative sample of the population of the area of Parma will be studied, divided on the basis of weight category, in order to assess water and salt intake and relationships with the presence of hypertension, and a sample of normal and hypertensive stone formers randomized to receive for one year either water therapy+low salt diet or water therapy alone.

DETAILED DESCRIPTION:
Background and rationale

Nephrolithiasis is a disease that could be defined as social, due to its widespread distribution and its continually increasing incidence in industrialized countries with a high standard of living (1). In Italy, it strikes just under 10% of the population, leading to expenditure of approx. 200 million euro/year for hospital admissions alone (2). Idiopathic Calcium Nephrolithiasis (ICN) with the formation of calcium oxalate stones, sometimes mixed with calcium phosphate ones, is the most common form, having an incidence of roughly 80% (3,4). As regards distribution in the two sexes, a slightly higher incidence in males has been observed. The pathogenesis of ICN involves both genetic and acquired factors (5), the combining of which leads to urinary biochemical anomalies which lie at the root of stone formation. A high rate of calcium-oxalate and/or calcium-phosphate supersaturation leads to the formation of nests of crystals that can then grow and aggregate to form a stone. The elements and urine compounds involved in the process of crystallization, whether they be inhibitors or promoters, are known as urinary stone risk factors. For Ca-oxalate they are: low urine volume (<2 l/day), hypercalciuria (>250mg/day), hyperoxaluria (>40 mg/day), hyperuricosuria (>600 mg/day), hypocitraturia (<320 mg/day) and hypomagnesuria (<50 mg/day). For Ca-phosphate, in addition to the above-mentioned factors, hyperphosphaturia (>1000 mg/day) and urinary pH also acquire considerable importance: a pH>7 promotes the formation of stones prevalently composed of phosphates, while a pH of between 6 and 7 associated with a urine volume <1l/day, can dangerously raise Ca-phosphate supersaturation and lead to the formation of mixed Ca-oxalate and Ca-phosphate stones. Finally, for uric acid stone disease the elements involved are hyperuricosuria and pH < 5.5. Among the stone risk factors, the most common found in the urine of patients affected by ICN is hypercalciuria with an incidence of around 50%. With regard to age of onset, there are two peaks, one between 20 and 30 years of age and one between 50 and 60.

Hypertension and obesity are also widespread social diseases with important epidemiological similarities to nephrolithiasis. These affinities have, over the years, led investigators to seek interconnections between the three diseases in order to find a common pathogenic moment. As far as hypertension is concerned, various studies have demonstrated that urinary excretion of calcium is greater in hypertensives than in normotensives. A linear association between the excretion of 24-h calcium and arterial blood pressure has been demonstrated in numerous studies, including INTERSALT (6). In 1999, after following up 132 hypertensives and 135 controls for 5 years, our group published a paper which reported the onset of stone disease in the hypertensives in significantly higher percentages compared to the controls, with an RR of 5.5 (7). Moreover, a year earlier, Madore and Curhan published two studies (8,9) conducted on a large cohort of Americans in which they demonstrated that patients with a past history of nephrolithiasis without hypertension were more prone to become hypertensive during the follow-up than non stone formers. These results, further confirmed by many subsequent studies, did not however succeed in clarifying the doubt as to whether it is the hypercalciuria of hypertensives that predisposes them to the development of stone disease or whether it is the renal damage, albeit microscopic, caused by stone disease that triggers the development of hypertension. Scientific literature has, however, identified, for hypertensives, stone formers and controls alike, a linear relationship between the excretion of calcium and the excretion of sodium, where calcium is the dependent variable and where the slope of the straight line, i.e. the increase of calcium for each mmol of sodium, is much greater in both stone formers and hypertensives than in controls. Moreover, as far back as the '80s, it was demonstrated that a reduction in kitchen salt intake from 10 g to 4 g per day, has the capacity to reduce calciuria more than a reduction in calcium intake from 1000 mg to 500 mg (10,11).

In 2002, we confirmed this experimental data with a paper published in the New England Journal of Medicine in which we demonstrated in recurrent male hypercalciuric stone formers followed up for 5 years, that a normal calcium, low-salt, low-protein diet had the power to reduce both the calciuria and the stone recurrences much more significantly than a low-calcium diet (12). Obviously it was not possible to separate the effect of the restriction of sodium from the restriction of protein. Both diets were accompanied by the recommendation to drink water, the effectiveness of which had already been demonstrated in first-episode stone formers in a previous study randomized with a follow-up of 5 years conducted on 199 stone formers and 101 controls (13).

The central role of body weight in determining stone risk is clearly described in scientific literature. BMI, weight, abdominal circumference are independently associated with kidney stone risk (14). Nevertheless, the mechanisms underlying this relation are still unknown. Data exist in literature to suggest that body weight can affect the excretion of many promoters or inhibitors of crystalline aggregation. For example, some population studies in the United States have demonstrated how urine pH is inversely correlated to body weight and how urinary excretion of calcium, oxalate and uric acid increase as body weight increases (15,16). Notwithstanding these data, the effects of body weight on the excretion of many urinary stone risk factors remains partly unknown; this is due to the limited weight categories, the low number of obese people in the study populations, the absence of a control group with "non stone formers" and the failure to record food intake in the studies published. In addition to this, as regards urinary excretion, the evaluation of excess weight solely on the basis of BMI values and abdominal circumference may seem somewhat reductive. It would appear to be more useful to assess body composition, lean mass, fat tissue mass and mineral mass. In this way, by better stratifying obesity classes, it might become simpler to understand the intricate endocrine/metabolic changes that occur in obesity (hyperinsulinism, hyperestrogenism etc.) and establish better correlations with the urinary excretion of stone risk factors. In fact, some studies (16) have demonstrated a slight increase in the total incidence of stone disease in female obese patients compared to males, with a slightly higher mean age in the females and, in any case, ages being equal, with a lower number of recurrences in the females compared to the males. These phenomena are probably affected by the concentration of serum estrogens and by the transformation in the fatty tissue of the adrenal androgens into estrogens; nonetheless the effects of serum estrogens on the urinary excretion of calcium are unknown. Finally, some studies have demonstrated that body weight also affects the composition of the stones. In fact, it has been demonstrated how the incidence of uric acid stones is higher in overweight/obese patients than in normal weight patients; some studies have highlighted that patients with idiopathic uric acid nephrolithiasis have a higher BMI than hyperuricosuric patients who form calcium oxalate stones. The pathophysiological link should be sought in hyperinsulinism: in fact insulin resistance is associated with a decrease in the production of renal ammonia leading to a consequent decrease in urinary pH, characteristic of uric acid stone disease (17). This theory is indirectly corroborated by the aforementioned indirect relationship between BMI and 24-h urine pH and the finding that also age-related reduced urinary acidification capacity increases the risk of uric stone disease, irrespective of body weight. On the basis of the above, it is clear how the presence of excess weight/obesity, uric acid or mixed stone disease could raise suspicions of a Metabolic Syndrome: there are, however, no conclusive studies on this, and neither have the effects on stone risk and arterial blood pressure of water therapy and a low-salt diet in a population of overweight/obese stone formers been sufficiently studied.

In the final analysis, nephrolithiasis, arterial hypertension and excess weight/obesity prove to be closely interconnected and it is possible to develop targeted diets aimed at reducing the risk of illness and death from this disease. Among such dietary approaches, the reduction of sodium chloride in food, increased hydration and an increased intake of foods with an alkaline potential (18) seem to play an important role.

For many years now, our research unit has been involved in projects, partially financed by the Italian Ministry of University and Research (MIUR), geared towards studying the effects induced by dietary changes in patients with calcium stone disease. The aim of the present project is to deepen our knowledge on the relationship between stone disease, hypertension, body weight and water and salt intake both in the general population of the area of Parma, where historically and by gastronomic tradition the normal diet tends to have a high salt content, and in a selected population of stone formers and hypertensives.

Experimental design/description of methodologies

As already mentioned, the aim of this project is to attempt to clarify the relationship between idiopathic calcium stone disease, salt and water intake, hypertension and body weight.

The study will be divided into two sub-projects:

1. Assessment of the salt and water intake in the general population of the area of Parma (duration 24 months)
2. Assessment of the effects of a low salt + water therapy diet vs water therapy alone for one year in patients with idiopathic calcium stone disease, both male and female, normal- and hypertensive without treatment (duration 12 months)

At least 350 healthy controls, 100 hypertensive non stone formers without treatment, 150 normotensive stone formers and 100 hypertensive stone formers without treatment will be enrolled in the study. Both the controls and the stone formers will be subdivided according to a 4-class BMI scale. The classes will have the following characteristics: Class 1 BMI £ 18.9 (underweight condition); Class 2 BMI between 19 and 24.9 (normal weight condition); Class 3 BMI between 25 and 29.9 (excess weight condition); Class 4 BMI > 30 (obesity). The patients enrolled will have their medical history recorded after which they will be subjected to the measurement of anthropometric parameters and arterial blood pressure, and a stone risk mini-profile will be drawn up including volume, creatinine, sodium, potassium and calcium measured according to the methods published. As is well-known, 24-h urinary sodium is considered the "gold standard" for the assessment of food-related salt intake, creatinine is a sensitive marker of lean mass, potassium is an index of the body's alkaline potential and calcium has the important pathophysiological role described above.

The stone formers will be randomized to receive a low salt+water therapy diet or water therapy alone, for one year. The term "water therapy" refers to an abundant intake of water with a low mineral and low sodium content (at least 2 litres in winter and 3 in summer). For stone formers only, at the end of the 12 month period of therapy, anthropometric parameters and arterial blood pressure will be measured once more and the urinary mini-profile will be repeated.

Objectives

Sub-project 1) "Assessment of the salt and water intake in the general population of the area of Parma"

Primary objective To assess the consumption of kitchen salt (NaCl) and the water intake in the general population of the area of Parma after adjustment for the BMI, and to study any possible relationships with the presence of arterial hypertension.

Secondary objectives

1. To study the urinary sodium-calcium relationship in the general normo- and hypertensive population without treatment.
2. To confirm the described relationship between 24-h calciuria and arterial blood pressure.
3. To identify any correlations between BMI and urinary solutes.
4. To stratify the salt and water intake by age category.
5. To assess the stone risk in the general normo- and hypertensive population without treatment.
6. To define urinary sodium-potassium-volume relationships in the general normo- and hypertensive population without treatment.

Sub-project 2) "Assessment of the effects of a low salt + water therapy diet vs water therapy alone for one year in patients with idiopathic calcium stone disease, both male and female, normal- and hypertensive without treatment (duration 12 months)"

Primary objective To assess the effects of a low-salt diet + water therapy vs water therapy alone, maintained for one year, on calciuria, arterial blood pressure and body weight in normo- and hypertensive stone formers.

Secondary objectives

1. To study the urinary sodium-calcium relationship in normo- and hypertensive stone formers without treatment and compare it with matched non stone formers.
2. To study the relationship between 24-h calciuria and arterial blood pressure in stone formers and compare it with matched non stone formers.
3. To identify any correlations between BMI and urinary solutes and evaluate the differences with matched non stone formers.
4. To stratify the salt and water intake by age category and recurrence rate in recurrent stone formers.
5. To assess the compliance with the low salt diet after one year.
6. To define the urinary sodium-potassium-volume relationships in normo- and hypertensive stone formers without treatment and compare them with matched non stone formers.

ELIGIBILITY:
For the stone formers main inclusion criteria

* age between 20 and 70 years
* caucasian race
* idiopathic calcium stone disease
* normal renal function (creatininemia <1.2 mg/dl)

Main exclusion criteria

* other major diseases
* diseases affecting the mineral and electrolyte metabolism (diabetes, endocrine diseases, inflammatory diseases etc.)
* treatments affecting the mineral and electrolytic metabolism (vitamin D, acetazolamide, anti-epilectic drugs, steroids etc).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
normalization of urinary stone risk factors | one year

SECONDARY OUTCOMES:
urinary sodium/calcium relationship | one yaer
blood pressure reduction | one year
relationship between 24h-calciuria and blood pressure | one year
stone rate reduction | one year
correlation BMI-urinary stone risk factors | one year
compliance | one year

CONTACTS AND LOCATIONS:
Overall Officials: Loris Borghi, Prof, Principal Investigator — University of Parma
Locations (1):
- University of Parma, Parma, Italy

REFERENCES:
- [Background] Goldfarb DS. Increasing prevalence of kidney stones in the United States. Kidney Int. 2003 May;63(5):1951-2. doi: 10.1046/j.1523-1755.2003.00942.x. No abstract available. PMID 12675877
- [Background] Elliott P, Stamler J, Nichols R, Dyer AR, Stamler R, Kesteloot H, Marmot M. Intersalt revisited: further analyses of 24 hour sodium excretion and blood pressure within and across populations. Intersalt Cooperative Research Group. BMJ. 1996 May 18;312(7041):1249-53. doi: 10.1136/bmj.312.7041.1249. PMID 8634612
- [Background] Goulding A, McParland BE. Fasting and 24-h urinary sodium/creatinine values in young and elderly women on low-salt and salt-supplemented regimens. J Cardiovasc Pharmacol. 1990;16 Suppl 7:S47-9. PMID 1708023
- [Background] Borghi L, Schianchi T, Meschi T, Guerra A, Allegri F, Maggiore U, Novarini A. Comparison of two diets for the prevention of recurrent stones in idiopathic hypercalciuria. N Engl J Med. 2002 Jan 10;346(2):77-84. doi: 10.1056/NEJMoa010369. PMID 11784873
- [Background] Taylor EN, Stampfer MJ, Curhan GC. Obesity, weight gain, and the risk of kidney stones. JAMA. 2005 Jan 26;293(4):455-62. doi: 10.1001/jama.293.4.455. PMID 15671430